CLINICAL TRIAL: NCT06189326
Title: Non-penetrating Deep Sclerectomy Versus Trabeculotomy- Trabeculectomy Operation in Treatment of Primary Congenital Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ehab Tharwat, Principal Investigator, Al-Azhar University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: primary congenital glaucoma
Record Dates: First submitted 2023-12-19; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Congenital Glaucoma
MeSH Terms: conditions — Hydrophthalmos

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-penetrating deep sclerectomy (Active Comparator)
  Interventions: Procedure: non-penetrating deep sclerectomy
- primary combined trabeculotomy-trabeculectomy (Active Comparator)
  Interventions: Procedure: primary combined trabeculotomy-trabeculectomy

INTERVENTIONS:
Procedure: non-penetrating deep sclerectomy — Non-penetrating deep sclerectomy (NPDS) is a non-perforating filtration procedure used for the surgical treatment of medically uncontrolled open angle glaucoma. This procedure was developed in an attempt to avoid many of the postoperative complications of trabeculectomy
  Arms: non-penetrating deep sclerectomy
Procedure: primary combined trabeculotomy-trabeculectomy — Combining trabeculotomy with trabeculectomy is one of the preferred surgical options, which showed favorable results in congenital glaucoma, and is advised mainly for treating moderate to severe forms of the disease, as the procedure provides dual pathways for aqueous drainage
  Arms: primary combined trabeculotomy-trabeculectomy

SUMMARY:
The high success rate of the non-penetrating deep sclerectomy (NPDS) procedure in adult glaucomatous patients motivated some glaucoma specialists to try it as an alternative procedure in childhood PCG. In deep sclerectomy, the surgeon fashions a partial-thickness scleral flap and excises the outer parts of both Schlemm's canal and trabecular meshwork without opening the eye, leaving a thin trabeculo-descemetic membrane. This membrane will guard against early postoperative hypotony due to the non-penetrating nature of the procedure.

The aim of this study is to assess the safety and efficacy outcomes of non-penetrating deep sclerectomy versus combined trabeculotomy-trabeculectomy in the treatment of congenital primary glaucoma

ELIGIBILITY:
Inclusion Criteria:

* patients with PCG younger than 6 years old with a HCD between 12-14 mm ware

Exclusion Criteria:

* patients with anterior segment anomalies,
* secondary glaucoma
* previous anterior segment surgeries
* patients more than 6 years old

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Intra Occular Pressure | Base line
  Intraocular pressure (IOP) is the fluid pressure of the eye. As pressure is a measure of force per area, IOP is a measurement involving the magnitude of the force exerted by the aqueous humor on the internal surface area of the anterior eye.
  It is measured by applanation tonometer its unite is mmHg
Intra Occular Pressure | Post 1 week
  Intraocular pressure (IOP) is the fluid pressure of the eye. As pressure is a measure of force per area, IOP is a measurement involving the magnitude of the force exerted by the aqueous humor on the internal surface area of the anterior eye.
  It is measured by applanation tonometer its unite is mmHg
Intra Occular Pressure | Post 1 month
  Intraocular pressure (IOP) is the fluid pressure of the eye. As pressure is a measure of force per area, IOP is a measurement involving the magnitude of the force exerted by the aqueous humor on the internal surface area of the anterior eye.
  It is measured by applanation tonometer its unite is mmHg
Intra Occular Pressure | Post 3 month
  Intraocular pressure (IOP) is the fluid pressure of the eye. As pressure is a measure of force per area, IOP is a measurement involving the magnitude of the force exerted by the aqueous humor on the internal surface area of the anterior eye.
  It is measured by applanation tonometer its unite is mmHg
Intra Occular Pressure | Post 6 month
  Intraocular pressure (IOP) is the fluid pressure of the eye. As pressure is a measure of force per area, IOP is a measurement involving the magnitude of the force exerted by the aqueous humor on the internal surface area of the anterior eye.
  It is measured by applanation tonometer its unite is mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Ehab tharwat, Damietta, New Damietta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided